CLINICAL TRIAL: NCT04178278
Title: The Reliability and Validity of Incremental Shuttle Walking Test to Assess Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Study for the Reliability and Validity of Incremental Shuttle Walking Test for COPD Patients in Korea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KOR-SWT
Record Dates: First submitted 2019-11-13; First posted 2019-11-26 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shuttle walking test group (Experimental): Patients will performed shultte walking test.
  Interventions: Diagnostic Test: Shuttle walking test
- Exercise stress test group (Active Comparator): Patients will performed exercise stress test.
  Interventions: Diagnostic Test: Exercise stress test
- 6 minutes walking test group (Active Comparator): Patients will performed 6 minutes walking test.
  Interventions: Diagnostic Test: 6 minutes walking test

INTERVENTIONS:
Diagnostic Test: Shuttle walking test — Patients will be required to walk around a 10-m course marked by cones placed 9 m apart, thus allowing 0.5 m for turning at each end. Walking speed will be regulated by prerecorded signals on a compact disc or MP3 file. Patients will increase walking speed at every minute. patients can stop this study, when they can not maintain their speeds due to dyspnea
  Arms: Shuttle walking test group
Diagnostic Test: Exercise stress test — Exercise stress test will be performed with cycle. When patients perform this study, they will gradually increase the velocity. Investigators will measure electrocardiography, vital sign, oxygen saturation, oxygen uptake, minute ventilation and fatigue.
  Arms: Exercise stress test group
Diagnostic Test: 6 minutes walking test — When participants perform 6 minutes walking test, patients will walk around the tract during 6 minutes. They can their walking speed according to condition and symptom. Investigators records walking distance, pulse rate, oxygen saturation and Borg scale
  Arms: 6 minutes walking test group

SUMMARY:
Investigators will perform this study to validate shuttle walking tests in korean patients with chronic obstructive pulmonary disease. This study will be performed as multi-center prospective observational correlation study in ulsan university hospital and asan medical center. 36 participants will perform the exercise stress test with cycle, 6 minutes walking test and shuttle walking test. Investigators will analyze correlation 6 minutes walking test and shuttle walking test with exercise stress test.

DETAILED DESCRIPTION:
Investigators will perform this study to validate shuttle walking tests in korean patients with chronic obstructive pulmonary disease. This study will be performed as multi-center prospective observational correlation study in ulsan university hospital and asan medical center.

18 patients will be enrolled in each hospital. When then visit, patients will perform questionnaire and laboratory study for baseline characteristics. After that, patients select memo, in which order for the exercise stress test with cycle, 6 minutes walking test and shuttle walking test will be written. Along that order, patients will perform each study at every two day in a week.

Investigators will analyze correlation 6 minutes walking test and shuttle walking test with exercise stress test. To analyze reliability in shuttle walking test, patients will shuttle walking test in two times. Researchers will analyze correlation between them.

ELIGIBILITY:
Inclusion Criteria:

* patients with respiratory symptom
* patients with forced expiratory volume 1/forced vital capacity < 0.7 in pulmonary function test after bronchodilator
* patients with informed consent

Exclusion Criteria:

* history of unstable angina or myocardial infarction within 1 month
* more than 120/mins pulse rate in stable state
* uncontrolled arrhythmia or history of syncope
* Symptomatic aortic stenosis or severe cardiac valve stenosis
* acute pulmonary embolism, deep vein thrombosis, aortic dissection or pulmonary edema
* difficult condition for shuttle walking test; visual, auditory or psychological disturbance
* respiratory failure
* oxygen saturation ≤ 85% in stable state
* needs for oxygen supply during walking
* active infection, acute infective endocarditis, renal failure, hyperthyroidism or significant pulmonary hypertension
* Left main coronary artery stenosis, hypertrophic cardiomyopathy
* systolic blood pressure more than 180 mmHg
* diastolic blood pressure more than 100 mmHg
* pregnant women
* patients with orthopedic disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between shuttle walking test, 6 minutes walking test and exercise stress test | 1 week
  Correlation between walking distance in shuttle walking test, walking distance in 6 minutes walking test and maximal oxygen uptake in exercise stress test

SECONDARY OUTCOMES:
Reproducibility in shuttle walking test | 1 week
  correlation between 2 times of walking distance in each shuttle walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpa, South Korea